CLINICAL TRIAL: NCT05484687
Title: Effect of Intravenous Infusion of Lidocaine on Patients Undergoing Radical Resection of Colorectal Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MA2021008
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Tumors; Lidocaine
Keywords: Radical resection of colorectal tumor; lidocaine; stress; immunity; vascular tumor regeneration; inflammation; micrometastasis
MeSH Terms: conditions — Colorectal Neoplasms; Inflammation; Neoplasm Micrometastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lidocaine is used in radical resection of colorectal tumors. (Experimental): Administer 1.5 mg/kg intravenously to the patient before induction of anesthesia, and continue to infuse 1.5 mg/kg/h during the operation until the end of the operation
  Interventions: Drug: Administer 1.5 mg/kg intravenously to the patient before induction of anesthesia, and continue to infuse 1.5 mg/kg/h during the operation until the end of the operation

INTERVENTIONS:
Drug: Administer 1.5 mg/kg intravenously to the patient before induction of anesthesia, and continue to infuse 1.5 mg/kg/h during the operation until the end of the operation — Administer 1.5 mg/kg lidocaine
  Other Names: same volume of saline

SUMMARY:
Colorectal cancer (CRC) is one of the most common malignant tumors in the world. Surgical resection is the main treatment option for colorectal cancer patients. Surgery may enhance or accelerate tumor recurrence and metastasis. Multiple factors in the tumor microenvironment play important roles in tumor recurrence and metastasis, and modulating the tumor microenvironment can inhibit disease progression. Lidocaine has been found to inhibit tumor growth in animal experiments.

DETAILED DESCRIPTION:
Lidocaine was applied in the operation of colorectal tumor patients, and the effect on the postoperative microenvironment and micrometastasis of the patients was observed by detecting the stress, immunity, vascular tumor regeneration, inflammation, etc. of the patients.

ELIGIBILITY:
Inclusion Criteria:

* colorectal tumor patients

Exclusion Criteria:

* Weight <45kg and >100kg
* Sensitivity or hypersensitivity to lidocaine
* Second or third degree heart block
* Severe heart failure (ejection fraction < 20%)
* History of active rhythm disorder
* Acute severe liver and kidney injury
* History of uncontrolled seizures
* History of acute porphyria.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
the concentration of tumor micrometastasis markers were determined by ELISA | 3 days after surgery
  the concentration of tumor micrometastasis markers such as CK20 was determined by ELISA

SECONDARY OUTCOMES:
the concentration of stress hormones were determined by ELISA | 3 days after surgery
  the concentration of EPI and NE were determined by ELISA
the concentration of inflammatory factor were determined by ELISA | 3 days after surgery
  the concentration of IL-6,IL-8,TNF-α were determined by ELISA
the concentration of angiogenesis factors were determined by ELISA | 3 days after surgery
  the concentration of VEGF was determined by ELISA
the concentration of immune indexes were determined by ELISA | 3 days after surgery
  the concentration of B lymphocytes, T lymphocytes, NK cells, macrophages were determined by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: hongsheng chen, Principal Investigator — Chair
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China